CLINICAL TRIAL: NCT01812759
Title: A Randomized Controlled Double-Blind Trial of Fentanyl Nasal Spray (Lazanda) Plus Hydromorphone Demand PCA Versus Placebo Nasal Spray Plus Hydromorphone Demand PCA for Treatment of Breakthrough Cancer Pain in the Emergency Department
Brief Title: Fentanyl for Breakthrough Pain in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Archimedes Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0982; NCI-2014-00915 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Pain
Keywords: Pain; Breakthrough cancer pain; Emergency Department; ED; Fentanyl nasal spray; Lazanda; Placebo nasal spray; Hydromorphone PCA; Dilaudid
MeSH Terms: conditions — Pain; Emergencies | interventions — Fentanyl; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fentanyl Nasal Spray + Hydromorphone PCA (Experimental): Fentanyl 100 mcg nasal spray administered plus hydromorphone PCA. All study patients receive demand dosing patient-controlled analgesia (PCA) with intravenous hydromorphone. Initial loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There will be no basal dose and the 8-hour dose limit will be 6.4 mg.
  Interventions: Drug: Fentanyl Nasal Spray; Drug: Hydromorphone PCA
- Placebo Nasal Spray + Hydromorphone PCA (Experimental): Placebo nasal spray administered plus hydromorphone PCA . All study patients receive demand dosing patient-controlled analgesia (PCA) with intravenous hydromorphone. Initial loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There will be no basal dose and the 8-hour dose limit will be 6.4 mg.
  Interventions: Drug: Hydromorphone PCA; Other: Placebo Nasal Spray

INTERVENTIONS:
Drug: Fentanyl Nasal Spray — 100 mcg nasal spray administered in each nostril.
  Other Names: Lazanda
  Arms: Fentanyl Nasal Spray + Hydromorphone PCA
Drug: Hydromorphone PCA — Initial loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There will be no basal dose and the 8-hour dose limit will be 6.4 mg.
  Other Names: Dilaudid
Other: Placebo Nasal Spray — 1 placebo nasal spray administered in each nostril.
  Arms: Placebo Nasal Spray + Hydromorphone PCA

SUMMARY:
The goal of this clinical research study is to learn if fentanyl nasal spray can help decrease pain related to cancer when used with other drugs for pain. Researchers also want to know if this drug can help decrease the length of your stay in the Emergency Department.

In this study, fentanyl nasal spray will be compared to a placebo nasal spray. A placebo is not a drug. It looks like the study drug but it is not designed to treat any disease or illness. It is designed in this study to be compared with the study spray to learn if the study spray has any real effect.

You will also be given intravenous (IV) pain drugs. You will be given these drugs even if you decide not to take part in this study.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to receive either fentanyl nasal spray or a placebo nasal spray. You will have an equal chance of being assigned to either group.

Neither you nor the study staff will know if you are receiving the study spray or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Visit and Study Treatment:

During your stay in the Emergency Department today, the following tests and procedures will be performed:

* Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be recorded.
* Information from your medical record about your age, sex, race, status of the disease, and any drugs that you may be taking for pain.
* The study nurse will also ask you some questions about your pain. It should take about 5 minutes to answer these questions.

You will then begin study treatment with either the fentanyl nasal spray or placebo nasal spray. The study nurse will help you use the nasal spray.

You will stay in the Emergency Department and will be monitored for up to 8 hours after the treatment has been administered. During this time, you will be asked about your pain and any side effects you may be having. The study nurse will also monitor your IV pain drug levels and other vital signs.

Length of Treatment:

Your active participation in this study will be over after your are monitored for up to 8 hours, at which time you will either be discharged to go home or admitted to the hospital based on your pain response and any other health problems that may be found during your visit to the Emergency Department.

Follow-Up Phone Call:

About 24 hours after your participation is over, the study nurse will call you by phone to ask if you experienced any other side effects since finishing the study treatment. The phone call should only last about 5 minutes. If you are still an inpatient at the hospital, the study nurse may visit you and ask you these questions in person.

This is an investigational study. Fentanyl nasal spray is FDA approved and commercially available for the treatment of pain. It's use to help with cancer pain in the Emergency Department is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients presenting to the Emergency Department for treatment of acute breakthrough pain who are already receiving and who are tolerant to opioid therapy for their underlying persistent cancer pain. (Patients considered opioid tolerant are those who are taking at least: 60 mg of oral morphine/day, 25 mcg of transdermal fentanyl/hour, 30 mg oral oxycodone/day, 8 mg oral hydromorphone/day, 25 mg oral oxymorphone/day, or an equianalgesic dose of another opioid for a week or longer.)
2. Patients must have severe pain on an 11-point Numeric Rating Scale (NRS 7-10)
3. Breakthrough cancer pain must be of sufficient severity to warrant the use of intravenous opioids in the judgment of the treating emergency physician
4. Age between 18 and 75 years
5. Able to understand the description of the study and give informed consent
6. Patients must be willing to and capable of providing frequent pain assessments for up to 8 hours
7. English-speaking

Exclusion Criteria:

1. Patients will not be approached while they are in acute distress and those exhibiting symptoms (such as dyspnea, uncontrolled nausea/vomiting or vertigo) to such an extent that impairs their ability to understand and evaluate informed consent
2. Patients participating in other clinical trials for pain
3. Patients who are not already tolerant to opioids
4. Patients, who in the judgment of the treating clinician, are suspected to have hepatic or renal failure
5. Patients who are pregnant or lactating
6. Patients with a known allergy or significant reaction to fentanyl, the components of the IN formulation, hydromorphone, or other opioids
7. Patients already on high morphine equivalent daily dose (MEDDs) (>500 mg/day).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2014-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knox H. Todd, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer patients presenting to the M. D. Anderson Cancer Center Emergency Department (ED) for treatment of acute breakthrough pain, who met study inclusion criteria.
Pre-assignment Details: The first patient's primary physician admitted the patient to the hospital after the patient consented to the study but before the patient received any medication.
Groups:
- Placebo: Placebo nasal spray administered in each nostril plus hydromorphone (PCA) Initial Patient Controlled Analgesia. (PCA) loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There was no basal dose and the 8-hour dose limit was 6.4 mg.
- Intervention: Fentanyl 100 mcg nasal spray administered in each nostril plus hydromorphone PCA. Initial PCA loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There was no basal dose and the 8-hour dose limit was 6.4 mg.
- No Medication: Patient consented but admitted to hospital before medication administered.
Period: Overall Study
Arm/Group | Placebo | Intervention | No Medication
Started | 1 | 1 | 1
Completed | 1 | 1 | 0
Not Completed | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo nasal spray administered in each nostril plus hydromorphone PCA. Initial PCA loading dose 0.2 mg with demand doses of 0.2 mg and lockout interval of 15 minutes. There was no basal dose and the 8-hour dose limit was 6.4 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | No Medication | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 1
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 3
Number of Participants with Pain Score between 7 and 10 using an 11- point (NRS) [Count of Participants; unit: Participants] — Pain Score between 7 and 10 using an 11-point National Rating Scale (NRS).The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
  Participants | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Total Pain Relief Score (TOTPAR4) at Four Hours After Treatment Initiation.
Description: Primary outcome is total pain relief score (TOTPAR4) at 4 hours after treatment initiation. TOTPAR4 defined as the sum of hourly pain relief scores after baseline to four hours after the first administered dose of Lazanda or placebo. Scores range from -1 (worse pain) to 4 (complete relief). Range of possible TOTPAR4 summed scores is -4 to 16. A TOTPAR4 score greater than or equal to 8 is considered a positive response.
Time Frame: 4 hours
Population: One participant consented but admitted to hospital before medication administered
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Intervention | No Medication
Number analyzed (Participants) | 1 | 1 | 0
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 11 Days
Arm/Group | Placebo | Intervention | No Medication
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes